CLINICAL TRIAL: NCT05571969
Title: A Phase Ib, Open Label, Multicenter Study to Determine the Maximum Tolerated Dose (MTD) of PARPi 2X-121 Monotherapy and the MTD of Dovitinib in Combination With 2X-121 in Patients With Advanced Solid Tumors
Brief Title: Study to Determine the Maximum Tolerated Dose (MTD) of PARPi 2X-121 Monotherapy and the MTD of Dovitinib in Combination With 2X-121 in Patients With Advanced Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Allarity Therapeutics (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-2003
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Intervention Model Description: This is a Phase Ib, two-part, multi-center study. In Part 1, the study will evaluate the safety and tolerability, antitumor activity, pharmacokinetics, and determine the maximum tolerated dose (MTD) of 2X-121 monotherapy (at BID regimen) in patients with advanced solid tumors. In Part 2, the study will evaluate the safety and tolerability, antitumor activity, and pharmacokinetics of 2X-121 (MTD) and dovitinib as combination therapy, and determine the MTD of dovitinib when given in combination with the MTD of 2X-121 determined in Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 2X-121 Monotherapy and Dovitinib in Combination with 2X-121 in Patients with Advanced Solid Tumors (Experimental): Determine the maximum tolerated dose (MTD) of 2X-121 monotherapy given twice daily (BID) and determine the MTD of dovitinib given in combination with 2X-121 (MTD) in patients with advanced solid tumors.
  Interventions: Drug: 2X-121 and dovitinib

INTERVENTIONS:
Drug: 2X-121 and dovitinib — The dose levels to be evaluated in Part 1 are:
  Cohort 1 600 mg (morning dose: 200 mg + evening dose: 400 mg); Cohort 2 800 mg (morning dose: 400 mg + evening dose: 400 mg); Cohort 3 1000 mg (morning dose: 400 mg + evening dose: 600 mg);
  The dose levels to be evaluated in Part 2 are:
  Cohort 1 2X-121 (MTD) + 300 mg dovitinib; Cohort 2 2X-121 (MTD) + 400 mg dovitinib; Cohort 3 2X-121 (MTD) + 500 mg dovitinib;

SUMMARY:
This is a Phase Ib, two-part, multi-center study. In Part 1, the study will evaluate the safety and tolerability, antitumor activity, pharmacokinetics, and determine the maximum tolerated dose (MTD) of 2X-121 monotherapy (at BID regimen) in patients with advanced solid tumors. In Part 2, the study will evaluate safety and tolerability, antitumor activity, pharmacokinetics and determine the MTD of dovitinib when given in combination with the MTD of 2X-121 determined in Part 1.

DETAILED DESCRIPTION:
Part 1

This part of the study will follow an accelerated titration method followed by a standard "3+3" design to determine the MTD of 2X-121. The MTD is defined as one dose level (cohort) below the dose in which dose limiting toxicities (DLTs) were observed in ≥ 33% of the participants.

The calculation of the sample size for this trial is based on the traditional 3 + 3 dose escalation scheme which is conducted as follows:

* Subjects are treated in cohorts of one (Cohort 1) or three (Cohorts 2-3) subjects, each receiving the same dose. For the assessment of a DLT, subjects are observed for 14 days.
* In Cohort 1, if the one subject does not exhibit a DLT, the next cohort of three subjects will receive the next higher dose (Cohort 2). In Cohort 2, if none of the three subjects exhibits a DLT, the next cohort of three subjects will receive the next higher dose (Cohort 3).
* Otherwise, if at least one subject of a cohort exhibits a DLT, a further cohort of three subjects is treated at the same dose level (cohort) without escalating the dose.
* If exactly one out of the six subjects treated at this dose exhibits a DLT, the trial continues as planned at the next higher dose level (cohort).
* If two or more subjects out of the six subjects treated at this dose exhibit a DLT, the dose escalation stops at that level and the next lower dose is considered as the MTD. When the escalation has stopped, additional subjects will be treated at the MTD to a total of six subjects.

Cohort escalation in Part 1 and Part 2 (i.e., the decision to progress from one cohort (dose level) to another) will not proceed until all of the following events have occurred:

1. All study subjects in a given cohort (dose level) have been enrolled, and
2. All such subjects have been followed for at least 14 days from the initiation of study treatment, and
3. The Investigator (PI), Sponsor's Medical Officer, and Medical Monitor have reviewed the available safety data, determined that none of the DLTs outlined below have occurred, and recommends further dose escalation

   * Hematological

     * Grade 4 neutropenia [or Grade 3 neutropenia with fever (>38.5 °C in axilla)] for ≥ 7 days
     * Grade 4 thrombocytopenia (Grade 3 thrombocytopenia with bleeding) lasting >7 days.
   * Other non-hematological toxicity

     * Grade 3 fatigue, or a 2-point decline in Eastern Cooperative Oncology Group (ECOG) performance status that persists for >7 days.
     * Nausea, vomiting or diarrhea that persists at Grade 3 or 4 despite maximal medical therapy.
     * Any Grade 3 or higher non-hematological laboratory abnormalities that require hospitalization.

The dose levels to be evaluated in Part 1 are shown below:

Cohort 1 600 mg (morning dose: 200 mg + evening dose: 400 mg)

Cohort 2 800 mg (morning dose: 400 mg + evening dose: 400 mg)

Cohort 3 1000 mg (morning dose: 400 mg + evening dose: 600 mg)

On Day 1 of first treatment cycle (C1D1), patients will be administered 2X-121 monotherapy as oral capsules taken twice daily. Each treatment cycle will consist of 28 days.

Blood samples will be collected for 2X-121 PK analysis at the following time points:

* C1D1: prior to drug administration (morning dose), 1 h (± 15 min), 3h (± 15 min), 4h (± 15 min), 6h (± 15 min), 12h (± 1 h, the sample should be taken before the evening dose)
* C1D2: prior to drug administration (morning dose)
* C1D7: prior to drug administration (morning dose)
* C1D15: prior to drug administration (morning dose)
* CXD1: prior to drug administration (morning dose) for the first day of all subsequent treatment cycles

Once the MTD has been determined, subjects enrolled in lower dose cohorts will be allowed to escalate the dose to the MTD, if acceptable per the Investigator's discretion. Subjects will be eligible for continuing treatment in absence of progressive disease or unacceptable toxicity or withdrawal of consent.

Part 2

In Part 2 of the study, patients will receive dovitinib in combination with the MTD of 2X-121 determined in Part 1. Part 2 will follow a "3+3" design to determine the MTD of dovitinib when given in combination with 2X-121. The MTD is defined as one dose level (cohort) below the dose in which dose limiting toxicities (DLTs) were observed in ≥ 33% of the participants. See Part 1 above for definition of DLTs.

The dose levels to be evaluated in Part 2 are shown below:

Cohort 1 2X-121 (MTD) + 300 mg dovitinib

Cohort 2 2X-121 (MTD) + 400 mg dovitinib

Cohort 3 2X-121 (MTD) + 500 mg dovitinib

Dovitinib will be administered once daily (morning) on a 5 days on/2 days off schedule. In a 28 day cycle, dovitinib will be administered C1D1 - C1D5, C1D8 - C1D12, C1D15 - C1D19, and C1D22 - C1D26.

Blood samples will be collected for 2X-121 and dovitinib PK analyses at the following time points:

* C1D1: prior to drug administration (morning dose), 0.5h (± 15 min), 1h (± 15 min), 2h (± 15 min), 3h (± 15 min), 4h (± 15 min), 6h (± 15 min), 8h (± 15 min), 10h (± 1 h), 12h (± 1 h, to be taken before the evening dose)
* C1D2: prior to drug administration (morning dose)
* C1D7: prior to drug administration (morning dose)
* C1D15: prior to drug administration (morning dose), 0.5h (± 15 min), 1h (± 15 min), 2h (± 15 min), 3h (± 15 min), 4h (± 15 min), 6h (± 15 min), 8h (± 15 min), 10h (± 1 h), 12h (± 1 h, to be taken before the evening dose)
* CXD1: prior to drug administration (morning dose) for the first day of all subsequent treatment cycles

Once the MTD has been determined, subjects enrolled in lower dose cohorts will be allowed to escalate the dose to the MTD, if acceptable per the Investigator's discretion. Subjects will be eligible for continuing treatment in absence of progressive disease or unacceptable toxicity or withdrawal of consent.

An additional 3-6 patients will receive 2X-121 in combination with dovitinib once the MTD dose is determined.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Histologically or cytological documented solid tumor.
3. Available tumor biopsy (most recent) for DRP® analysis.
4. Measurable disease by CT scan or MRI if possible.
5. Performance status of ECOG ≤ 1.
6. Recovered to Grade <1 or baseline from prior surgery or from acute toxicities of prior radiotherapy, or from treatment with cytotoxic, hormonal or biologic agents.
7. ≥ 2 weeks must have elapsed since any prior surgery or therapy with G-CSF and GM-CSF.
8. Patients with intracranial disease must be on stable or decreased level of steroid therapy (e.g. dexamethasone) for at least 7 days prior to baseline MRI. Non-enzymatic inducing anti-epileptic drugs are allowed.
9. Adequate conditions as evidenced by the following clinical laboratory values:

   1. Absolute neutrophils count (ANC) ≥ 1500/mm3 (1.5 x 10³/mL)
   2. Hemoglobin > 10.0 g/dL
   3. Platelets ≥ 100,000/mm3 (≥ 100 x 10⁹/L)
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN or ≤5x ULN in presence of liver metastases
   5. Serum bilirubin ≤ 1.5 ULN
   6. Alkaline phosphatase ≤ 2.5 x ULN
   7. Creatinine ≤ 1.5 ULN
   8. Blood urea nitrogen (BUN) ≤2X ULN.
10. Life expectancy equal or longer than 3 months.
11. The subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided and has had the opportunity to discuss the study with the investigator or designee.
12. The subject is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
13. The subject is able to understand the nature of the study and any potential hazards associated with participating in it.
14. Negative pregnancy test for female subjects of childbearing potential. Women of childbearing potential (WOCBP) and Women of non-childbearing potential are eligible to participate. Both women of childbearing potential and women of non-childbearing potential should use an approved method of birth control and agree to continue to use this method for the duration of the study (and for 90 days after taking the last dose of study drug).

Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only) (e.g., diaphragm, cervical cap, male condom, and female condom and spermicidal foam, sponges, and film), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile for at least three months before screening or 2 years post-menopausal at time of screening. All male subjects/partners must agree to consistently and correctly use a condom for the duration of the study and for 90 days after taking the study drug. In addition, subjects may not donate sperm for the duration of the study and for 90 days after taking study drug.

-

Exclusion Criteria:

1. Concurrent chemotherapy, radiotherapy, hormonal therapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period.
2. Other malignancy with exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to entering the study.
3. Any active infection requiring parenteral or oral antibiotic treatment.
4. History of coagulation or bleeding disorder or subject currently on therapeutic anticoagulant medication.

   Note: Prophylactic doses of heparin or low molecular weight heparin are allowed.
5. Known HIV positivity.
6. Known active hepatitis B or C.
7. Clinically significant (i.e. active) cardiovascular disease:

   1. Stroke within ≤ 6 months prior to day 1
   2. Transient ischemic attack (TIA) within ≤ 6 months prior to day 1
   3. Myocardial infarction within ≤ 6 months prior to day 1
   4. Unstable angina
   5. New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF)
   6. Serious cardiac arrhythmia requiring medication.
8. Other medications or conditions, including surgery, that in the Investigator's opinion would contraindicate study participation for safety reasons or interfere with the interpretation of study results.
9. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of 2X-121 and dovitinib.
10. Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
11. Female patients who are pregnant or breast-feeding (pregnancy test with a positive result before study entry).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the MTD of 2X-121 monotherapy. | Evaluated after up to approximately 2 years
  To determine the maximum tolerated dose (MTD) of 2X-121 monotherapy given twice daily (BID) in patients with advanced solid tumors.
Determination of the MTD of dovitinib given in combination with 2X-121 (MTD). | Evaluated after up to approximately 2 years
  To determine the MTD of dovitinib given in combination with 2X-121 (MTD) in patients with advanced solid tumors.

SECONDARY OUTCOMES:
To evaluate the objective response rate (ORR) of 2X-121 monotherapy (Part 1) and in combination with dovitinib (Part 2). | Evaluated after up to approximately 2 years
  ORR is defined as the proportion of subjects who achieve a Complete Response (CR) or Partial Response (PR) as assessed by RECIST v1.1.
To evaluate the duration of overall response (DOR) of 2X-121 monotherapy (Part 1) and in combination with dovitinib (Part 2). | Evaluated after up to approximately 2 years
  DOR is defined as the time in months from the first documented CR or PR per RECIST v. 1.1 to disease recurrence or disease progression (PD) whichever occurs first.
To evaluate progression free survival (PFS) of 2X-121 monotherapy (Part 1) and in combination with dovitinib (Part 2). | Evaluated after up to approximately 2 years
  PFS is defined as the time from study treatment initiation to either first observation of progressive disease or occurrence of death.
To evaluate overall survival (OS) of 2X-121 monotherapy (Part 1) and in combination with dovitinib (Part 2). | Evaluated after up to approximately 2 years
  OS is defined as the time from study treatment initiation to death from any cause or last day known to be alive.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Carolina BioOncology, Huntersville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio